CLINICAL TRIAL: NCT05630430
Title: The Effect of Volar Carbon Plate Applications on Radiation Exposure and Procedure Time in Intra-articular Radius Distal End Fractures
Brief Title: Volar Carbon Plate Effects on Procedure Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed Cagatay Engin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-03-29; First posted 2022-11-29 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Radiation Exposure; Surgery; Radius Distal Fracture
Keywords: carbon plate; radius distal; radiation; surgery
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volar Carbon Plate Effects on Procedure Time (Experimental): Carbon alloy plates, offer the advantage of faster radiological reduction control because they do not create superposition to the fracture line
  Interventions: Procedure: The Effect of Volar Carbon Plate Applications on Radiation Exposure and Procedure Time in Intra-articular Radius Distal End Fractures
- Titanium Alloy Plates Group (Active Comparator): Titanium alloy plates are frequently used materials in our current orthopedic surgery practices. The main goal during surgical treatment is to obtain an accurate and acceptable bone alignment. Since titanium alloy plates are radiopaque, they create a superposition to the fracture line and more than one view is usually required in each plane to ensure the reduction quality during surgery.
  Interventions: Procedure: The Effect of Volar Carbon Plate Applications on Radiation Exposure and Procedure Time in Intra-articular Radius Distal End Fractures

INTERVENTIONS:
Procedure: The Effect of Volar Carbon Plate Applications on Radiation Exposure and Procedure Time in Intra-articular Radius Distal End Fractures — Surgery procedure, Although the bones are at the surgeon's disposal in plate fixation of radius distal end fractures, fluoroscopy is frequently used for reduction control. The increase in the need for scopy both directly affects the duration of the operation and causes the surgical team to be exposed to excessive radiation. Since titanium alloy plates are radiopaque, they create a superposition to the fracture line and more than one view is usually required in each plane to ensure the reduction quality during surgery. Carbon alloy plates, on the other hand, offer the advantage of faster radiological reduction control because they do not create superposition to the fracture line. In our study, in addition to the comparisons in the literature, it is aimed to investigate the effect of carbon plates on the procedure time. surgery time and exposure of radiation will be recorded at the end of the surgery
  Other Names: Titanium Alloy Plate surgery; Carbon Alloy Plate surgery

SUMMARY:
Radius distal end fractures are common orthopedic injuries. Many methods have been described in the treatment of distal radius fractures. The fixation of radius distal end fracture with volar plate was first applied by Ellis in 1965. Over the years, ideas have been put forward on the materials used for plates and the radiolucent carbon fiber plates has been used. These plates cause less artifact in computed tomography (CT) and magnetic resonance examinations (MRI), allow a better evaluation of the fracture, exhibit biomechanical characteristics close to the cortical bone, and do not cause a coldwedding in patients.

DETAILED DESCRIPTION:
Titanium alloy plates are frequently used materials in our current orthopedic surgery practices. The main goal during surgical treatment is to obtain an accurate and acceptable bone alignment. Achieving this goal as soon as possible will reduce additional morbidity and mortality and increase the success of treatment. Therefore, studies aiming to reduce the operation time come to the fore. When the literature is examined, there are limited number of studies on carbon plates. In these studies, it was reported that similar functional results were obtained with titanium alloy plates. Although the bones are at the surgeon's disposal in plate fixation of radius distal end fractures, fluoroscopy is frequently used for reduction control. The increase in the need for scopy both directly affects the duration of the operation and causes the surgical team to be exposed to excessive radiation. Since titanium alloy plates are radiopaque, they create a superposition to the fracture line and more than one view is usually required in each plane to ensure the reduction quality during surgery. Carbon alloy plates, on the other hand, offer the advantage of faster radiological reduction control because they do not create superposition to the fracture line. In our study, in addition to the comparisons in the literature, it is aimed to investigate the effect of carbon plates on the procedure time. For this purpose, distal radius fractured patients applied to our clinic will be treated with titanium and carbon plates after the necessary randomization. After the tourniquet is applied, the time elapsed until the fixation is completed, the duration of scopy, and the number of scopy images taken will be recorded. In the follow-ups, the functional scores and radiological measurements of the patients will be made and the complications will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Radius distal simple intraarticular fractures
* Closed fractures

Exclusion Criteria:

* Acompanying fracture at the same limb
* Open fractures
* Pathological fractures
* The patients who don't want to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Procedures Time | 0-1 hours of the surgery
  Time elapsed in minutes between the starting of the surgical procedure and the fixation time.
Radiation Exposure | 0-1 hours of the surgery
  Time elapsed in minutes during the surgery
Functional Outcome | At the end of the 2nd week
  wrist flexion degree measurement with goniometer , wrist extension degree measurement with goniometer , ulnar deviation degree measurement with goniometer and radial deviation degree measurement with goniometer and measurement with a hand grip strength dynamometer
Functional Outcome | At the end of the 5th week
  wrist flexion degree measurement with goniometer , wrist extension degree measurement with goniometer , ulnar deviation degree measurement with goniometer and radial deviation degree measurement with goniometer and measurement with a hand grip strength dynamometer
Functional Outcome | At the end of the 3rd month
  wrist flexion, extension, ulnar deviation and radial deviation degree measurement with wrist flexion degree measurement with goniometer , wrist extension degree measurement with goniometer , ulnar deviation degree measurement with goniometer and radial deviation degree measurement with goniometer and measurement with a hand grip strength dynamometer
Functional Outcome | At the end of the 6th month
  wrist flexion degree measurement with goniometer , wrist extension degree measurement with goniometer , ulnar deviation degree measurement with goniometer and radial deviation degree measurement with goniometer and measurement with a hand grip strength dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No